CLINICAL TRIAL: NCT02185755
Title: Investigating if an Internet-Based Glucose Monitoring System is as Effective as Medication at Reducing HbA1c Levels in Type 2 Diabetes Mellitus
Brief Title: Internet Monitoring vs Medication to Control Blood Sugar in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, ERS Gap Student, Medical Director, Endocrine Research Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IBGMS standalone
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Internet-Based Glucose Monitoring System; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-Based Glucose Monitoring System (Active Comparator): The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and provide feedback limited to non-medicine related comments and suggestions.
  Interventions: Other: Internet-Based Glucose Monitoring System
- Normal Medication Positive Control (Other): The subjects will be prescribed a new medication as appropriate for normal therapy. This group will receive no biweekly feedback nor require to report online, but will see the endocrinologist every 3 months up to 6 months.
  Interventions: Drug: Normal Medication Positive Control

INTERVENTIONS:
Other: Internet-Based Glucose Monitoring System
  Other Names: Internet Blood Glucose Monitoring System; Remote Blood Glucose Monitoring System
  Arms: Internet-Based Glucose Monitoring System
Drug: Normal Medication Positive Control
  Arms: Normal Medication Positive Control

SUMMARY:
Managing blood sugar levels is important for patients with type 2 diabetes (T2DM) to minimize health problems and complications. One way for patients to notify doctors and receive feedback about their blood sugar management is through an online system. As Internet-based glucose monitoring systems (IBGMS) have already been shown to be effective, the investigators hypothesize that IBGMS is effective as an intervention even when limiting feedback to non-medicine related changes.

DETAILED DESCRIPTION:
1. Purpose:

   To determine the effectiveness of an Internet-based glucose monitoring system (IBGMS) in the absence of medication changes.
2. Hypothesis:

   IBGMS without medication changes is comparable to conventional medication at reducing HbA1c levels over 8% in patients with T2DM.
3. Justification:

   Patients with T2DM having elevated HbA1c levels may be prescribed additional medications to help manage their blood sugar levels, which include oral hypoglycemic agents and/or insulin. As IBGMS has been shown to be effective in reducing HbA1c in T2DM, there is an opportunity to determine whether if this system could be used as an alternative to medication.

   The benefits would include reduced side effects as a result of substituting for the effects of medication, as well as reduced financial costs associated with acquiring medication.

   Considering that IBGMS increases the frequency at which patients receive feedback to change medications as compared to typical treatment, the risk is as typical for a patient opting for no medication changes for the same period of time.
4. Objectives: The primary end-point is to determine if patients using IBGMS have reduced HbA1c values at followup, and to compare the reduction to the control group on typical medications.
5. Research Method: 120 patients with T2DM satisfying the inclusion criteria will be recruited and have baseline HbA1c established through regular lab blood tests. They will be randomized into one of two groups, one that will be trained to use IBGMS and one control group going on an appropriate additional medication.

   The IBGMS group will be asked to report their blood sugars to their endocrinologist biweekly and receive feedback for each report. No medication changes will be offered in the feedback, but lifestyle or dietary recommendations may be included.

   The control group will be asked to take their new medications as indicated by their endocrinologist.

   Both groups will have followup visits with their endocrinologist at 3 and 6 months, and will also have blood tests done at those time points checking their HbA1c levels.

   The effectiveness of both interventions will be evaluated individually and against each other.

   For the IBGMS group, a rescue secondary endpoint occurs if a subject maintains an HbA1c level at or greater than 8% after 3 months; the subject will be withdrawn from the study and put under standard care.
6. Statistical Analysis: The sample size was calculated to be 120 by estimating mean differences and standard deviations using data from previous studies. For the calculation the statistical power was 0.80 and alpha of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients being treated with oral hypoglycemic agents
* HbA1c > 8%
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be trained on using the Internet-Based Glucose Monitoring System
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet access on a computer
* No prior use or training on IBGMS

Exclusion Criteria:

* Patient with medical conditions that may affect their study participation or results will be excluded.
* Patients using medications known to influence control of diabetes (eg steroids systemic or inhaled)
* Liver disease (AST (aspartate aminotransferase) or ALT (alanine aminotransferase) levels > 2.5 times the reference level)
* Renal insufficient with a serum creatinine level > 200 μmol/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
HbA1c Levels before and after intervention | 6 months
  Compare HbA1c Levels before and after intervention for both arms, as well as the difference in HbA1c Levels between arms.

SECONDARY OUTCOMES:
The secondary endpoint include severe hypoglycemia defined as requiring external aid (hospital or other). | 6 months
A secondary endpoint includes adverse events such as unplanned hospitalizations for any cause that last more than 24 hours | 6 months
HbA1c levels remain at 8% or higher | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh D Tildesley, MD, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- Dr. Hugh Tildesley Inc., Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] Tildesley HD, Mazanderani AB, Ross SA. Effect of Internet therapeutic intervention on A1C levels in patients with type 2 diabetes treated with insulin. Diabetes Care. 2010 Aug;33(8):1738-40. doi: 10.2337/dc09-2256. PMID 20668152
- [Background] Cho JH, Chang SA, Kwon HS, Choi YH, Ko SH, Moon SD, Yoo SJ, Song KH, Son HS, Kim HS, Lee WC, Cha BY, Son HY, Yoon KH. Long-term effect of the Internet-based glucose monitoring system on HbA1c reduction and glucose stability: a 30-month follow-up study for diabetes management with a ubiquitous medical care system. Diabetes Care. 2006 Dec;29(12):2625-31. doi: 10.2337/dc05-2371. PMID 17130195